CLINICAL TRIAL: NCT04236323
Title: The Effect of Remifentanil on Rebound Pain in Patients Receiving General Anesthesia for Shoulder Arthroplasty After Brachial Plexus Block for Postoperative Pain Control
Brief Title: The Effect of Remifentanil on Rebound Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1912-041-1087
Record Dates: First submitted 2020-01-15; First posted 2020-01-22 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Pain, Postoperative
Keywords: hyperalgesia; brachial plexus block; remifentanil
MeSH Terms: conditions — Pain, Postoperative; Hyperalgesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- not used intraoperative remifentanil infusion (Experimental): Adult patients aged < 70 years and ASA class < III undergoing rotator cuff repair not used intraoperative remifentanil infusion
  Interventions: Drug: Not used remifentanil infusion
- used intraoperative remifentanil infusion (No Intervention): Adult patients aged < 70 years and ASA class < III undergoing rotator cuff repair used intraoperative remifentanil infusion maintaining target concentration of 2-6ng/ml

INTERVENTIONS:
Drug: Not used remifentanil infusion — Remifentanil is not used during operation
  Arms: not used intraoperative remifentanil infusion

SUMMARY:
The investigators will evaluate the influence of intraoperative remifentanil infusion on the postoperative hyperalgesia in patients receiving rotator cuff repair after brachial plexus block for postoperative analgesia.

DETAILED DESCRIPTION:
The study will include 68 patients undergoing rotator cuff repair. All patients will receive brachial plexus block for postoperative analgesia, followed by general anesthesia. In the experimental group, remifentanil infusion will not be used intraoperatively, and in the control group, remifentanil will be infused. After surgery, both groups will be given the same postoperative pain management using patient controlled analgesia(PCA), and pain patterns will be assessed using the Numerical rating scale (NRS) at 4 hour intervals for 24 hours. The primary end point of this study is the total dose of PCA medication over 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I,II,III
* Patients undergoing arthroscopic rotator cuff repair surgery under general anesthesia after interscalen brachial plexus block for post operative analgesia
* Age ranges from 20 to 70

Exclusion Criteria:

* Patients who didn't agree to study
* Patients can't control PCA(Patient-Controlled-Analgesia) independently
* Patients who have conciousness disorder or can't express their pain level by NRS(Numeric Rating Scale) system
* Patients who have severe respiratory disease or hepatic failure
* Patinets who have known neuropathy or coagulopathy
* Pregnancy
* Patients with allegies to the drugs used in this study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Total infused dose of patient controlled analgesia(PCA) drug during 24 hours | From end of operation to the 24hours after operation
  Total infused dose of patient controlled analgesia(PCA) drug during first 24 hours after rotor cuff repair under general anesthesia

SECONDARY OUTCOMES:
Numerical Ratings Scale | Pain levels are checked using Numerical Ratings Scale at 4 hour intervals for 24 hours after surgery
  Degree of pain is assessed using Numerical Ratings Scale at 4 hours for 24 hours after operation. The patients choose one of the digits from 0 to 10, the zero-point is painless, and the ten-point means the one with the most severe pain.
Total patient's trial to PCA bolus infusion | 24 hours after surgery
  The total number of times patients press the infusion button on the PCA to control pain
Incidence of postoperative nausea and vomiting | 24 hours after surgery
  Postoperative nausea and vomiting is assessed at 24hr after surgery by a face-to face interview

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD., PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No